CLINICAL TRIAL: NCT02942277
Title: Phase 1 Dose Escalating, Double-Blind, Randomized Comparator Controlled Trial of the Safety andImmunogenicity of Pfs25M-EPA/AS01 and Pfs230D1M-EPA/AS01 Vaccines, Transmission Blocking Vaccines Against Plasmodium Falciparum at Full and Fractional Dosing in Adults in Mali
Brief Title: Safety and Immunogenicity of Pfs25M-EPA/AS01 and Pfs230D1M-EPA/AS01 Vaccines, Transmission Blocking Vaccines Against Plasmodium Falciparum, at Full and Fractional Dosing in Adults in Mali
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 999917006; 17-I-N006
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Results first posted 2022-01-28 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2020-07-29

CONDITIONS: Malaria
Keywords: Malaria; Reactogenicity; Antibody; Direct Skin Feed; Mosquito
MeSH Terms: conditions — Malaria | interventions — Engerix-B; Meningococcal Vaccines; Saline Solution; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- 1a (Experimental): (n=5), to receive 16 microgram Pfs25M-EPA/AS01 on D0, D28, D168
  Interventions: Biological: Pfs25M-EPA; Other: AS01; Other: Normal Saline
- 1b (Experimental): (n=10), to receive 47 microgram Pfs25M-EPA/AS01 on D0, D28, D168
  Interventions: Biological: Pfs25M-EPA; Other: AS01
- 2a (Experimental): (n=5), to receive 13 microgram Pfs230D1M-EPA/AS01 on D0, D28, D168
  Interventions: Biological: Pfs230D1M-EPA; Other: AS01; Other: Normal Saline
- 2b (Experimental): (n=10), to receive 40 microgram Pfs230D1M-EPA/AS01 on D0, D28, D168
  Interventions: Biological: Pfs230D1M-EPA; Other: AS01
- 2c (Experimental): (n=60), to receive 40 micrograms Pfs230D1M-EPA/AS01 on D0, D28, D168; all subjects will undergo antimalarial drug treatment with Coartem on D-7 (prior to vaccination #1); 4th vaccination on D476
  Interventions: Biological: Pfs230D1M-EPA; Other: AS01; Drug: Coartem
- 2d (Experimental): (n=60), to receive 40 micrograms Pfs230D1M-EPA/AS01 (500 (Micro)L TBV + AS01) on D0, D28, then 8 micro liters Pfs230D1M- EPA/AS01 (100 (Micro)L TBV + AS01;fractional dose) on D168; all subjects will undergo antimalarial drug treatment with Coartem on D-7 (prior to vaccination #1); 4th vaccination on D476
  Interventions: Biological: Pfs230D1M-EPA; Other: AS01; Drug: Coartem
- 3a (Experimental): (n=5), to receive 16 microgram Pfs25M-EPA/AS01 and 13 microgram Pfs230D1M-EPA/AS01 on D0, D28, D168
  Interventions: Biological: Pfs25M-EPA; Biological: Pfs230D1M-EPA; Other: AS01; Other: Normal Saline
- 3b (Experimental): (n=10), to receive 47 microgram Pfs25M-EPA/AS01 and 40 microgram Pfs230D1M-EPA/AS01 on D0, D28, D168 (Bamako)
  Interventions: Biological: Pfs25M-EPA; Biological: Pfs230D1M-EPA; Other: AS01
- 4a (Active Comparator): (n=10), to receive ENGERIX-B on D0, D28, and D168
  Interventions: Biological: Engerix-B; Other: Normal Saline
- 4b (Active Comparator): (n=10), to receive ENGERIX-B on DO, D28, and Dl68
  Interventions: Biological: Engerix-B; Drug: Coartem
- 4c (Active Comparator): (n=120), to receive ENGERIX-B on D0, D28, and D168 (start study with Arm 2c and 2d); all subjects will undergo antimalarial drug treatment with Coartem on D-7 (prior to vaccination #1); vaccination with Menactra on D476
  Interventions: Biological: Engerix-B; Biological: Menactra; Drug: Coartem

INTERVENTIONS:
Biological: Pfs25M-EPA — The PpPfs25M and EcEPA lots, both manufactured at Walter Reed Bioproduction facility (Silver Spring, Maryland) in cGMP compliance, were used to manufacture the conjugate. PpPfs25M is a Pichia- expressed recombinant Pfs25 with a molecular mass of 18,713 Daltons.The Pfs25M- EPA was formulated as conjugated Pfs25M in 4 mM PBS to a 2X dilution of the high dose (188 (Micro)g/ml in 0.5 ml volume) in cGMP compliance at Walter Reed Bio-production facility in April 2016 and will be provided as a single use vial.
  Arms: 1a; 1b; 3a; 3b
Biological: Pfs230D1M-EPA — The Pfs230D1M-EPA was formulated as conjugated Pfs230D1M in 4 mM PBS to a 2X dilution of the high dose (160 (Micro)g/ml in 0.5 ml volume) in cGMP compliance at Walter Reed Bio-production facility in April 2016 and will be provided as a single use vial.
  Arms: 2a; 2b; 2c; 2d; 3a; 3b
Other: AS01 — AS01B adjuvant will also be provided as a single use vial by GSK, 100 microgram/mL MPL and 100microgram/mL QS21 in a liposomal formulation in a volume of 0.625 mL. One dose injected of AS01B corresponds to 50 μg QS21 and 50 μg MPL.
  Arms: 1a; 1b; 2a; 2b; 2c; 2d; 3a; 3b
Biological: Engerix-B — ENGERIX-B (hepatitis B vaccine; recombinant): is a sterile suspension of noninfectious hepatitis B virus surface antigen (HBsAg) for intramuscular administration. It contains purified HBsAg obtained by culturing genetically engineered Saccharomyces cerevisiae cells, which carry the surface antigen gene of the hepatitis B virus. Each 1-mL adult dose contains 20 g of HBsAg adsorbed on 0.5 mg aluminum as aluminum hydroxide. FDA approved for persons 20 years of age and older for a series of 3 doses on a 0-, 1-, 6-month schedule.
  Arms: 4a; 4b; 4c
Biological: Menactra — Menactra is FDA approved for active immunization to prevent invasive meningococcal disease caused by Neisseria meningitidis serogroups A, C, Y, and W-135 (but does not protect against serotype B) for use in individuals 9 months through 55 years of age
  Arms: 4c
Other: Normal Saline — Sterile isotonic (0.9%) normal saline will be commercially procured in the US and shipped to Mali at ambient temperature. Normal saline will be administered in a 0.5 mL dose as an intramuscular injection. Normal saline will also be used for diluting Pfs25M-EPA and Pfs230D1M-EPA prior to formulation with AS01B for the lower dose groups in Bamako, Mali.
  Arms: 1a; 2a; 3a; 4a
Drug: Coartem — Artemether/lumefantrine (Coartem(R)) is a licensed antimalarial in the US and Mali for treatment of uncomplicated malaria. It has an excellent safety profile and is widely used to treat malaria. Subjects who may have any contraindications to the use of these drugs will be excluded at screening. Coartem will be dosed with food and administered over 3 days for a total of 6 doses, as per package insert and standard adult dosing
  Arms: 2c; 2d; 4b; 4c

SUMMARY:
Background:

Researchers are looking for new ways to control and eradicate malaria. They want to test vaccines to block malaria transmission in adults in Mali. These vaccines work by inducing antibodies in a person. The antibody is then taken up with blood by a mosquito that bites the person. This blocks parasite development in the mosquito. This stops malaria transmission to another person.

Objective:

To test the safety, reactogenicity, immunogenicity, and transmission-blocking activity of the vaccines Pfs25M-EPA and Pfs230D1M-EPA with AS01 in Malian adults.

Eligibility:

Healthy Malians ages 18-50 living in certain areas in Mali who:

Are not pregnant or breastfeeding

Are not infected with HIV, Hepatitis B and Hepatitis C

Do not have evidence of immunodeficiency

Do not have history of severe allergic reaction or anaphylaxis

Design:

Participants will be screened with:

Medical history

Physical exam

Malaria Comprehension Exam

Blood and urine tests

Electrocardiogram (for participants in certain study groups)

Participants will be randomly assigned to a study group.

Participants will be monitored for 12-16 months. For the first 7 months, they will have between 1 and nine visits a month. The number depends on the month and on what group they are in. For the rest of the months, they will have 1 monthly visit.

Each visit includes a physical exam. Most include blood tests.

Participants will get 3 doses of a study or comparator vaccine. They get the vaccine through an injection in the upper arm. This occurs at their first visit, then 1 month later, and then 5 months later.

Participants will be followed for at least 6 months after the last vaccine.

If participants develop an injection site rash or reaction, photographs may be taken of the site.

DETAILED DESCRIPTION:
A vaccine to interrupt malaria transmission (VIMT) would be a valuable tool for local elimination or eradication of this disease, and may contain components that block transmission to mosquitoes (such as Pfs25 or Pfs230) or that prevent human infection (such as the vaccine RTS,S). Pfs25 and Pfs230, surface antigens of zygotes and ookinetes (and gametocytes for Pfs230) in the mosquito stage of P. falciparum, are the lead candidates for a malaria transmission blocking vaccine (TBV). Recombinant Pfs25M and recombinant Pfs230D1M have each been conjugated to P. aeruginosa ExoProtein A (EPA) and adjuvanted with AS01. Our ongoing experience with Pfs25M-EPA and Pfs230D1M-EPA in Malian adult trial participants, and the extensive experience with the AS01 adjuvants in African children and adults, justify conducting the first-in-human trial of Pfs25M-EPA and Pfs230D1M-EPA with AS01 in Malian adults. This dose-escalating phase 1 study will determine safety, immunogenicity, and functional activity of these vaccines in Malian adults. Pfs25M-EPA + Pfs230D1M-EPA in AS01 will be assessed by mosquito feeding assays in Malian adults for evidence that they may reduce the number of malaria transmission events in study subjects.

A total of 305 subjects will be enrolled at multiple sites in Mali, West Africa to receive escalating doses of a malaria transmission blocking vaccine (s): Pfs25M-EPA/AS01, Pfs230D1M-EPA/AS01, or simultaneous administration of Pfs25M-EPA/AS01 and Pfs230D1M-EPA/AS01; or a comparator vaccine (ENERGIX-B). Enrollment within each group will be staggered for additional safety and subjects will only be enrolled into the co-administration group once each individual dose has been administered. Subjects will be followed for at least 6 months after the last vaccination. Safety outcomes will be local and systemic adverse events and serious adverse events. Immunogenicity outcomes will be antibody responses as measured by ELISA against recombinant Pfs25, Pfs230, EPA, CSP, and B cell and T cell responses. Functional activity of the induced antibodies will be assessed in TBV arms by standard membrane feeding assays conducted at the National Institute of Allergy and Infectious Diseases, and activity that interrupts malaria transmission will be measured in all arms by direct skin feeding assays in Mali.

Subjects in the open label safety cohorts (Arms 1a, 1b, 2a, 2b, 3a, 3b, 4a, 4b) will be offered reenrollment for follow-up laboratory assessment to explore the duration of immunogenicity and functional activity at approximately 9, 12 months post vaccination. Following scheduled, intentional unblinding, subjects enrolled in Arms 2c, 2d, and 4c will be provided the opportunity to re-enroll for a fourth vaccination (Arm 2c and 2d with 40 microgram dose of Pfs230D1M-EPA/AS01; Arm 4c with Menatctra) approximately 1 year post vaccination #3. Subjects in these arms will also be eligible to re-enroll for follow up of duration of immunogenicity and functional activity at approximately 9, 12 months post vaccination if they choose not to enroll to recive the booster vaccination. Subjects will be followed similarly to the previous year for safety, immunogenicity, and functional activity.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Age greater than or equal to 18 and less than or equal to 50 years.
2. Available for the duration of the trial.
3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
4. In good general health and without clinically significant medical history in the opinion of the investigator.
5. Females of childbearing potential must be willing to use reliable contraception (as defined below) from 21 days prior to Study Day 0 (Study Day 476 for re-enrollment) and then until 3 months after last vaccination.

   * Reliable methods of birth control include one of the following: confirmed pharmacologic contraceptives (parenteral) delivery; intrauterine or implantable device.
   * Reliable methods of birth control include concurrent use of a pharmacologic and a barrier method, i.e. two of the following: confirmed pharmacologic contraceptives (oral, transdermal) delivery or vaginal ring AND condoms with spermicide or diaphragm with spermicide.
   * Non-childbearing women will also be required to report date of last menstrual period, history of surgical sterility (i.e. tubal ligation, hysterectomy) or premature ovarian insufficiency (POI), and will have a baseline urine or serum pregnancy test performed.
6. Willingness to have blood samples stored for future research.
7. Willingness to undergo DSFs (Arms 3c, 3d, 4c only).
8. Known resident of Bancoumana or Doneguebougou or surrounding area or known student or long term resident (more than 1 year) of Bamako/Sotuba, Mali

EXCLUSION CRITERIA:

1. Pregnancy as determined by a positive urine or serum human choriogonadotropin (beta-hCG) test (if female).

   NOTE: Pregnancy is also a criteria for discontinuation of any further dosing or non-safety related interventions for that subject.
2. Currently breast-feeding (if female).
3. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and comply with the study protocol.
4. Hemoglobin, WBC, absolute neutrophils, and platelets outside the local laboratory-defined limits of normal (subjects may be included at the investigator s discretion for not clinically significant values outside of normal range and less than or equal to Grade 1).
5. Alanine transaminase (ALT) or creatinine (Cr) level above the local laboratory-defined upper limit of normal (subjects may be included at the investigator s discretion for not clinically significant values outside of normal range and less than or equal to Grade 1).
6. Infected with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B (HBV).
7. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies including urinalysis.
8. History of receiving any investigational product within the past 30 days.
9. Participation or planned participation in a clinical trial with an investigational product prior to completion of the follow up visit 28 days following last vaccination OR planned participation in an investigational vaccine study until the last required protocol visit
10. Subject has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
11. History of a severe allergic reaction or anaphylaxis.
12. Severe asthma, defined as asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past 2 years, or that has required the use of oral or parenteral corticosteroids at any time during the past 2 years.
13. Pre-existing autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sj(SqrRoot)(Delta)gren s syndrome, or autoimmune thrombocytopenia.
14. Known immunodeficiency syndrome.
15. Known asplenia or functional asplenia.
16. Use of chronic (greater than or equal to 14 days) oral or intravenous corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone >10 mg/day) or immunosuppressive drugs within 30 days of Study Day 0.
17. Prior to Study Day 0 and every subsequent vaccination day, receipt of a live vaccine within the past 4 weeks or a killed vaccine within the past 2 weeks.
18. Receipt of immunoglobulins and/or blood products within the past 6 months.
19. Previous receipt of an investigational malaria vaccine in the last 5 years.
20. History of severe reaction to mosquito bites (Arms 3c, 3d, 4c only)
21. History of allergy to the comparator vaccine (such as latex, yeast, or previous Hepatitis B vaccine)
22. Known allergies or contraindications (such as significant cardiac disease; prolonged QTc >450 ms; currently taking medications that may prolong your QTc; serious side effects from Coartem in the past) to study treatment (Coartem [artemether/lumefantrine]) (Arms 3c, 3d, 4c only)
23. Other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant participating in the trial, interfere with the evaluation of the study objectives, or would render the subject unable to comply with the protocol.

Ages: 18 Years to 52 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 301 (Actual)
Dates: Start 2016-10-21; Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick E Duffy, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Bancoumana Malaria Vaccine Center, Bamako, Mali

REFERENCES:
- [Background] Wu Y, Przysiecki C, Flanagan E, Bello-Irizarry SN, Ionescu R, Muratova O, Dobrescu G, Lambert L, Keister D, Rippeon Y, Long CA, Shi L, Caulfield M, Shaw A, Saul A, Shiver J, Miller LH. Sustained high-titer antibody responses induced by conjugating a malarial vaccine candidate to outer-membrane protein complex. Proc Natl Acad Sci U S A. 2006 Nov 28;103(48):18243-8. doi: 10.1073/pnas.0608545103. Epub 2006 Nov 16. PMID 17110440
- [Background] Tachibana M, Wu Y, Iriko H, Muratova O, MacDonald NJ, Sattabongkot J, Takeo S, Otsuki H, Torii M, Tsuboi T. N-terminal prodomain of Pfs230 synthesized using a cell-free system is sufficient to induce complement-dependent malaria transmission-blocking activity. Clin Vaccine Immunol. 2011 Aug;18(8):1343-50. doi: 10.1128/CVI.05104-11. Epub 2011 Jun 29. PMID 21715579
- [Background] Diallo M, Toure AM, Traore SF, Niare O, Kassambara L, Konare A, Coulibaly M, Bagayogo M, Beier JC, Sakai RK, Toure YT, Doumbo OK. Evaluation and optimization of membrane feeding compared to direct feeding as an assay for infectivity. Malar J. 2008 Dec 2;7:248. doi: 10.1186/1475-2875-7-248. PMID 19055715
- [Derived] Healy SA, Sagara I, Assadou MH, Katile A, Kone M, Imeru A, Kwan JL, Swihart BJ, Fintzi J, Potter GE, Zeguime A, Dolo A, Diarra B, Narum DL, Rausch KM, MacDonald NJ, Zhu D, Mohan R, Thera I, Morrison RD, Zaidi I, Doritchamou JYA, Sylla D, Hume JCC, Coulibaly MB, Morelle D, Lievens M, Doumbo OK, Duffy PE; Pfs230D1 Vaccine Team. A Vaccine to Block Plasmodium falciparum Transmission. NEJM Evid. 2025 Jul;4(7):EVIDoa2400188. doi: 10.1056/EVIDoa2400188. Epub 2025 Jun 24. PMID 40552966
- [Derived] Cao Y, da Silva Araujo M, Lorang CG, Dos Santos NAC, Tripathi A, Vinetz J, Kumar N. Distinct immunogenicity outcomes of DNA vaccines encoding malaria transmission-blocking vaccine target antigens Pfs230D1M and Pvs230D1. Vaccine. 2025 Feb 15;47:126696. doi: 10.1016/j.vaccine.2024.126696. Epub 2025 Jan 8. PMID 39787798

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Community permission was obtained from village elders and other community members in Sotuba/Bamako, Bancoumana, and Doneguebougou after explanation and discussion of the study at a community meeting. A general announcement inviting household and family members to the participating clinic to learn about the study was made at the time of community permission, using local radio or any traditional channel of communication.
Groups:
- Pilot/Safety Arm 1a: Dosing Interval 0, 28, 168 Days: Participants received 3 doses of 16 μg Pfs25M-EPA/AS01 via intramuscular injections into the deltoid muscle (IM) on D0, D28, D168
  Pfs25M-EPA: The PpPfs25M and EcEPA lots, both manufactured at Walter Reed Bioproduction facility (Silver Spring, Maryland) in cGMP compliance, were used to manufacture the conjugate. PpPfs25M is a Pichia- expressed recombinant Pfs25 with a molecular mass of 18,713 Daltons.
  The Pfs25M- EPA was formulated as conjugated Pfs25M in 4 mM PBS to a 2X dilution of the high dose (188 μg/ml in 0.5 ml volume) in cGMP compliance at Walter Reed Bio-production facility in April 2016 and provided as a single use vial.
  AS01: AS01B adjuvant was provided as a single use vial by GSK, 100 μg/mL MPL and 100 μg/mL QS21 in a liposomal formulation in a volume of 0.625 mL. One dose injected of AS01B corresponds to 50 μg QS21 and 50 μg MPL.
  Normal Saline: Sterile isotonic (0.9%) normal saline was commercially procured in the US and shipped to Mali at ambient temperature. Normal saline was administered in a 0.5 mL dose as an intramuscular injection. Normal saline was also used for diluting Pfs25M-EPA and Pfs230D1M-EPA prior to formulation with AS01B for the lower dose groups in Bamako, Mali.
- Pilot/Safety Arm 1b: Dosing Interval 0, 28, 168 Days: Participants received 3 doses of 47 μg Pfs25M-EPA/AS01 via intramuscular injections into the deltoid muscle (IM) on D0, D28, D168
  Pfs25M-EPA: The PpPfs25M and EcEPA lots, both manufactured at Walter Reed Bioproduction facility (Silver Spring, Maryland) in cGMP compliance, were used to manufacture the conjugate. PpPfs25M is a Pichia- expressed recombinant Pfs25 with a molecular mass of 18,713 Daltons.
  The Pfs25M- EPA was formulated as conjugated Pfs25M in 4 mM PBS to a 2X dilution of the high dose (188 μg/ml in 0.5 ml volume) in cGMP compliance at Walter Reed Bio-production facility in April 2016 and was provided as a single use vial.
  AS01: AS01B adjuvant was provided as a single use vial by GSK, 100 μg/mL MPL and 100 μg/mL QS21 in a liposomal formulation in a volume of 0.625 mL. One dose injected of AS01B corresponds to 50 μg QS21 and 50 μg MPL.
- Pilot/Safety Arm 2a: Dosing Interval 0, 28, 168 Days: Participants received 3 doses of 13 μg Pfs230D1M-EPA/AS01 via intramuscular injections into the deltoid muscle (IM) on D0, D28, D168
  Pfs230D1M-EPA: The Pfs230D1M-EPA was formulated as conjugated Pfs230D1M in 4 mM PBS to a 2X dilution of the high dose (160 μg/ml in 0.5 ml volume) in cGMP compliance at Walter Reed Bio-production facility in April 2016 and was provided as a single use vial.
  AS01: AS01B adjuvant was provided as a single use vial by GSK, 100 μg/mL MPL and 100 μg/mL QS21 in a liposomal formulation in a volume of 0.625 mL. One dose injected of AS01B corresponds to 50 μg QS21 and 50 μg MPL.
  Normal Saline: Sterile isotonic (0.9%) normal saline was commercially procured in the US and shipped to Mali at ambient temperature. Normal saline was administered in a 0.5 mL dose as an intramuscular injection. Normal saline was used for diluting Pfs25M-EPA and Pfs230D1M-EPA prior to formulation with AS01B for the lower dose groups in Bamako, Mali.
- Pilot/Safety Arm 2b: Dosing Interval 0, 28, 168 Days: Participants received 3 doses of 40 μg Pfs230D1M-EPA/AS01 via intramuscular injections into the deltoid muscle (IM) on D0, D28, D168
  Pfs230D1M-EPA: The Pfs230D1M-EPA was formulated as conjugated Pfs230D1M in 4 mM PBS to a 2X dilution of the high dose (160 μg/ml in 0.5 ml volume) in cGMP compliance at Walter Reed Bio-production facility in April 2016 and was provided as a single use vial.
  AS01: AS01B adjuvant was provided as a single use vial by GSK, 100 μg/mL MPL and 100 μg/mL QS21 in a liposomal formulation in a volume of 0.625 mL. One dose injected of AS01B corresponds to 50 μg QS21 and 50 μg MPL.
- Safety/Efficacy Arm 2c: Dosing Interval 0, 28, 168, 476 Days: Participants received 3 doses of 40 μg Pfs230D1M-EPA/AS01 via intramuscular injections into the deltoid muscle (IM) on Days 0, 28, 168, and a 4th dose on Day 476 (Year 2). Participants received antimalarial drug treatment with Coartem® approximately 1 week prior to first vaccination.
  Pfs230D1M-EPA: The Pfs230D1M-EPA was formulated as conjugated Pfs230D1M in 4 mM PBS to a 2X dilution of the high dose (160 (Micro)g/ml in 0.5 ml volume) in cGMP compliance at Walter Reed Bio-production facility in April 2016 and was provided as a single use vial.
  AS01: AS01B adjuvant was provided as a single use vial by GSK, 100 μg/mL MPL and 100 μg/mL QS21 in a liposomal formulation in a volume of 0.625 mL. One dose injected of AS01B corresponds to 50 μg QS21 and 50 μg MPL.
  Coartem: Artemether/lumefantrine (Coartem(R)) is a licensed antimalarial in the US and Mali for treatment of uncomplicated malaria. It has an excellent safety profile and is widely used to treat malaria. Subjects who may have had any contraindications to the use of these drugs were excluded at screening. Coartem was dosed with food and administered over 3 days for a total of 6 doses, as per package insert and standard adult dosing
- Safety/Efficacy Arm 2d: Dosing Interval 0, 28, 168, 476 Days: Participants received 3 doses of 40 μg Pfs230D1M-EPA/AS01 on Days 0, 28, then 8 μg Pfs230D1M-EPA/AS01 (100 µL TBV + AS01; fractional dose) on Day 168, then 4th dose of 40 μg Pfs230D1M-EPA/AS01 on Day 476 (Year 2) via intramuscular injections into the deltoid muscle (IM). Participants received antimalarial drug treatment with Coartem® approximately 1 week prior to first vaccination.
  Participants underwent antimalarial drug treatment with Coartem on D-7 (prior to vaccination #1); 4th vaccination on D476
  Pfs230D1M-EPA: The Pfs230D1M-EPA was formulated as conjugated Pfs230D1M in 4 mM PBS to a 2X dilution of the high dose (160 μg/ml in 0.5 ml volume) in cGMP compliance at Walter Reed Bio-production facility in April 2016 and was provided as a single use vial.
  AS01: AS01B adjuvant was provided as a single use vial by GSK, 100 μg/mL MPL and 100 μg/mL QS21 in a liposomal formulation in a volume of 0.625 mL. One dose injected of AS01B corresponds to 50 μg QS21 and 50 μg MPL.
  Coartem: Artemether/lumefantrine (Coartem(R)) is a licensed antimalarial in the US and Mali for treatment of uncomplicated malaria. It has an excellent safety profile and is widely used to treat malaria. Subjects who may have had any contraindications to the use of these drugs were excluded at screening. Coartem was dosed with food and administered over 3 days for a total of 6 doses, as per package insert and standard adult dosing
- Pilot/Safety Arm 3a: Dosing Interval 0, 28, 168 Days: Participants received 3 doses of 16 μg Pfs25M-EPA/AS01 and 13 μg Pfs230D1M-EPA/AS01 via intramuscular injections into the deltoid muscle (IM) on Days 0, 28, 168
  Pfs25M-EPA: The PpPfs25M and EcEPA lots, both manufactured at Walter Reed Bioproduction facility (WRB; Silver Spring, Maryland) in cGMP compliance, were used to manufacture the conjugate. PpPfs25M is a Pichia-expressed recombinant Pfs25 with a molecular mass of 18,713 Daltons. The Pfs25M-EPA was formulated as conjugated Pfs25M in 4 mM PBS to a 2X dilution of the high dose (188 μg/ml in 0.5 ml volume) in cGMP compliance at WRB facility in Apr 2016 and was provided as a single use vial.
  Pfs230D1M-EPA: The Pfs230D1M-EPA was formulated as conjugated Pfs230D1M in 4 mM PBS to a 2X dilution of the high dose (160 μg/ml in 0.5 ml volume) in cGMP compliance at Walter Reed Bio-production facility in April 2016 and was provided as a single use vial.
  AS01: AS01B adjuvant was provided as a single use vial by GSK, 100 μg/mL MPL and 100 μg/mL QS21 in a liposomal formulation in a volume of 0.625 mL. One dose injected of AS01B corresponds to 50 μg QS21 and 50 μg MPL.
  Normal Saline: Sterile isotonic (0.9%) normal saline will be commercially procured in the US and shipped to Mali at ambient temperature. Normal saline was administered in a 0.5 mL dose as an intramuscular injection. Normal saline was be used for diluting Pfs25M-EPA and Pfs230D1M-EPA prior to formulation with AS01B for the lower dose groups in Bamako, Mali.
- Pilot/Safety Arm 3b: Dosing Interval 0, 28, 168 Days: Participants received 3 doses of 47 μg Pfs25M-EPA/AS01 and 40 μg Pfs230D1M-EPA/AS01 via intramuscular injections into the deltoid muscle (IM) on Days 0, 28, 168
  Pfs25M-EPA: The PpPfs25M and EcEPA lots, both manufactured at Walter Reed Bioproduction facility (Silver Spring, Maryland) in cGMP compliance, were used to manufacture the conjugate. PpPfs25M is a Pichia-expressed recombinant Pfs25 with a molecular mass of 18,713 Daltons. The Pfs25M-EPA was formulated as conjugated Pfs25M in 4 mM PBS to a 2X dilution of the high dose (188 μg/ml in 0.5 ml volume) in cGMP compliance at Walter Reed Bio-production facility in April 2016 and was provided as a single use vial.
  Pfs230D1M-EPA: The Pfs230D1M-EPA was formulated as conjugated Pfs230D1M in 4 mM PBS to a 2X dilution of the high dose (160 μg/ml in 0.5 ml volume) in cGMP compliance at Walter Reed Bio-production facility in April 2016 and was provided as a single use vial.
  AS01: AS01B adjuvant was provided as a single use vial by GSK, 100 μg/mL MPL and 100 μg/mL QS21 in a liposomal formulation in a volume of 0.625 mL. One dose injected of AS01B corresponds to 50 μg QS21 and 50 μg MPL.
- Pilot/Safety Comparator Arm 4a: Dosing Interval 0, 28, 168 Days: Participants received 3 doses of ENGERIX-B via intramuscular injections into the deltoid muscle (IM) on Days 0, 28, and 168
  Engerix-B: ENGERIX-B (hepatitis B vaccine; recombinant): is a sterile suspension of noninfectious hepatitis B virus surface antigen (HBsAg) for intramuscular administration. It contains purified HBsAg obtained by culturing genetically engineered Saccharomyces cerevisiae cells, which carry the surface antigen gene of the hepatitis B virus. Each 1-mL adult dose contains 20 g of HBsAg adsorbed on 0.5 mg aluminum as aluminum hydroxide. FDA approved for persons 20 years of age and older for a series of 3 doses on a 0-, 1-, 6-month schedule.
  Normal Saline: Sterile isotonic (0.9%) normal saline was commercially procured in the US and shipped to Mali at ambient temperature. Normal saline was administered in a 0.5 mL dose as an intramuscular injection. Normal saline was also used for diluting Pfs25M-EPA and Pfs230D1M-EPA prior to formulation with AS01B for the lower dose groups in Bamako, Mali.
- Pilot/Safety Comparator Arm 4b: Dosing Interval 0, 28, 168 Days: Participants received 3 doses of ENGERIX-B via intramuscular injections into the deltoid muscle (IM) on Days 0, 28, and 168
  Engerix-B: ENGERIX-B (hepatitis B vaccine; recombinant): is a sterile suspension of noninfectious hepatitis B virus surface antigen (HBsAg) for intramuscular administration. It contains purified HBsAg obtained by culturing genetically engineered Saccharomyces cerevisiae cells, which carry the surface antigen gene of the hepatitis B virus. Each 1-mL adult dose contains 20 g of HBsAg adsorbed on 0.5 mg aluminum as aluminum hydroxide. FDA approved for persons 20 years of age and older for a series of 3 doses on a 0-, 1-, 6-month schedule.
  Coartem: Artemether/lumefantrine (Coartem(R)) is a licensed antimalarial in the US and Mali for treatment of uncomplicated malaria. It has an excellent safety profile and is widely used to treat malaria. Subjects who may have had any contraindications to the use of these drugs were excluded at screening. Coartem was dosed with food and administered over 3 days for a total of 6 doses, as per package insert and standard adult dosing
- Safety Comparator & Efficacy Comparator Arm 4c: Dosing Interval 0, 28, 168, 476 Days: Participants received 3 doses of ENGERIX-B via on Days 0, 28, and 168, then 4th vaccination of Menactra® on Day 476 (Year 2) via intramuscular injections into the deltoid muscle (IM). Participants received antimalarial drug treatment with Coartem® approximately 1 week prior to first vaccination.
  Engerix-B: ENGERIX-B (hepatitis B vaccine; recombinant): is a sterile suspension of noninfectious hepatitis B virus surface antigen (HBsAg) for intramuscular administration. It contains purified HBsAg obtained by culturing genetically engineered Saccharomyces cerevisiae cells, which carry the surface antigen gene of the hepatitis B virus. Each 1-mL adult dose contains 20 g of HBsAg adsorbed on 0.5 mg aluminum as aluminum hydroxide.
  Menactra: Menactra is FDA approved for active immunization to prevent invasive meningococcal disease caused by Neisseria meningitidis serogroups A, C, Y, and W-135 (but does not protect against serotype B) for use in individuals 9 months through 55 years of age
  Coartem: Artemether/lumefantrine (Coartem®) is a licensed antimalarial in the US and Mali for treatment of uncomplicated malaria. It has an excellent safety profile and is widely used to treat malaria. Subjects who may have had any contraindications to the use of these drugs were excluded at screening. Coartem was dosed with food and administered over 3 days for a total of 6 doses, as per package insert and standard adult dosing
Period: Year 1
Arm/Group | Pilot/Safety Arm 1a: Dosing Interval 0, 28, 168 Days | Pilot/Safety Arm 1b: Dosing Interval 0, 28, 168 Days | Pilot/Safety Arm 2a: Dosing Interval 0, 28, 168 Days | Pilot/Safety Arm 2b: Dosing Interval 0, 28, 168 Days | Safety/Efficacy Arm 2c: Dosing Interval 0, 28, 168, 476 Days | Safety/Efficacy Arm 2d: Dosing Interval 0, 28, 168, 476 Days | Pilot/Safety Arm 3a: Dosing Interval 0, 28, 168 Days | Pilot/Safety Arm 3b: Dosing Interval 0, 28, 168 Days | Pilot/Safety Comparator Arm 4a: Dosing Interval 0, 28, 168 Days | Pilot/Safety Comparator Arm 4b: Dosing Interval 0, 28, 168 Days | Safety Comparator & Efficacy Comparator Arm 4c: Dosing Interval 0, 28, 168, 476 Days
Started | 5 | 10 | 5 | 10 | 56 | 61 | 5 | 10 | 10 | 10 | 119
Completed | 5 | 8 | 5 | 9 | 49 | 51 | 5 | 9 | 10 | 10 | 104
Not Completed | 0 | 2 | 0 | 1 | 7 | 10 | 0 | 1 | 0 | 0 | 15
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 3
Not completed — Travel | 0 | 1 | 0 | 0 | 4 | 5 | 0 | 0 | 0 | 0 | 8
Not completed — Joined Army | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject met withdrawal criteria | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Year 2
Arm/Group | Pilot/Safety Arm 1a: Dosing Interval 0, 28, 168 Days | Pilot/Safety Arm 1b: Dosing Interval 0, 28, 168 Days | Pilot/Safety Arm 2a: Dosing Interval 0, 28, 168 Days | Pilot/Safety Arm 2b: Dosing Interval 0, 28, 168 Days | Safety/Efficacy Arm 2c: Dosing Interval 0, 28, 168, 476 Days | Safety/Efficacy Arm 2d: Dosing Interval 0, 28, 168, 476 Days | Pilot/Safety Arm 3a: Dosing Interval 0, 28, 168 Days | Pilot/Safety Arm 3b: Dosing Interval 0, 28, 168 Days | Pilot/Safety Comparator Arm 4a: Dosing Interval 0, 28, 168 Days | Pilot/Safety Comparator Arm 4b: Dosing Interval 0, 28, 168 Days | Safety Comparator & Efficacy Comparator Arm 4c: Dosing Interval 0, 28, 168, 476 Days
Started | 5 | 8 | 5 | 9 | 49 | 51 | 5 | 9 | 10 | 10 | 104
Completed | 5 | 7 | 4 | 8 | 36 | 40 | 4 | 8 | 10 | 9 | 79
Not Completed | 0 | 1 | 1 | 1 | 13 | 11 | 1 | 1 | 0 | 1 | 25
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Did not rescreen | 0 | 0 | 1 | 1 | 9 | 6 | 0 | 1 | 0 | 0 | 21
Not completed — Met withdrawal criteria | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1
Not completed — Travel | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3
Not completed — Non-compliant | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pilot/Safety Arm 1a: Dosing Interval 0, 28, 168 Days: Participants received 3 doses of 16 μg Pfs25M-EPA/AS01 via intramuscular injections into the deltoid muscle (IM) on D0, D28, D168
- Pilot/Safety Arm 1b: Dosing Interval 0, 28, 168 Days: Participants received 3 doses of 47 μg Pfs25M-EPA/AS01 via intramuscular injections into the deltoid muscle (IM) on D0, D28, D168
- Pilot/Safety Arm 2a: Dosing Interval 0, 28, 168 Days: Participants received 3 doses of 13 μg Pfs230D1M-EPA/AS01 via intramuscular injections into the deltoid muscle (IM) on D0, D28, D168
- Pilot/Safety Arm 2b: Dosing Interval 0, 28, 168 Days: Participants received 3 doses of 40 μg Pfs230D1M-EPA/AS01 via intramuscular injections into the deltoid muscle (IM) on D0, D28, D168
- Safety/Efficacy Arm 2c: Dosing Interval 0, 28, 168, 476 Days: Participants received 3 doses of 40 μg Pfs230D1M-EPA/AS01 via intramuscular injections into the deltoid muscle (IM) on Days 0, 28, 168, and a 4th dose on Day 476 (Year 2). Participants received antimalarial drug treatment with Coartem® approximately 1 week prior to first vaccination.
- Safety/Efficacy Arm 2d: Dosing Interval 0, 28, 168, 476 Days: Participants received 3 doses of 40 μg Pfs230D1M-EPA/AS01 on Days 0, 28, then 8 μg Pfs230D1M-EPA/AS01 (100 µL TBV + AS01; fractional dose) on Day 168, then 4th dose of 40 μg Pfs230D1M-EPA/AS01 on Day 476 (Year 2) via intramuscular injections into the deltoid muscle (IM). Participants received antimalarial drug treatment with Coartem® approximately 1 week prior to first vaccination.
- Pilot/Safety Arm 3a: Dosing Interval 0, 28, 168 Days: Participants received 3 doses of 16 μg Pfs25M-EPA/AS01 and 13 μg Pfs230D1M-EPA/AS01 via intramuscular injections into the deltoid muscle (IM) on Days 0, 28, 168
- Pilot/Safety Arm 3b: Dosing Interval 0, 28, 168 Days: Participants received 3 doses of 47 μg Pfs25M-EPA/AS01 and 40 μg Pfs230D1M-EPA/AS01 via intramuscular injections into the deltoid muscle (IM) on Days 0, 28, 168
- Pilot/Safety Comparator Arm 4a: Dosing Interval 0, 28, 168 Days; Pilot/Safety Comparator Arm 4b: Dosing Interval 0, 28, 168 Days: Participants received 3 doses of ENGERIX-B via intramuscular injections into the deltoid muscle (IM) on Days 0, 28, and 168
- Safety Comparator & Efficacy Comparator Arm 4c: Dosing Interval 0, 28, 168, 476 Days: Participants received 3 doses of ENGERIX-B via on Days 0, 28, and 168, then 4th vaccination of Menactra® on Day 476 (Year 2) via intramuscular injections into the deltoid muscle (IM). Participants received antimalarial drug treatment with Coartem® approximately 1 week prior to first vaccination.
- Total: Total of all reporting groups
Arm/Group | Pilot/Safety Arm 1a: Dosing Interval 0, 28, 168 Days | Pilot/Safety Arm 1b: Dosing Interval 0, 28, 168 Days | Pilot/Safety Arm 2a: Dosing Interval 0, 28, 168 Days | Pilot/Safety Arm 2b: Dosing Interval 0, 28, 168 Days | Safety/Efficacy Arm 2c: Dosing Interval 0, 28, 168, 476 Days | Safety/Efficacy Arm 2d: Dosing Interval 0, 28, 168, 476 Days | Pilot/Safety Arm 3a: Dosing Interval 0, 28, 168 Days | Pilot/Safety Arm 3b: Dosing Interval 0, 28, 168 Days | Pilot/Safety Comparator Arm 4a: Dosing Interval 0, 28, 168 Days | Pilot/Safety Comparator Arm 4b: Dosing Interval 0, 28, 168 Days | Safety Comparator & Efficacy Comparator Arm 4c: Dosing Interval 0, 28, 168, 476 Days | Total
Number analyzed (Participants) | 5 | 10 | 5 | 10 | 56 | 61 | 5 | 10 | 10 | 10 | 119 | 301
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 10 | 5 | 10 | 56 | 61 | 5 | 10 | 10 | 10 | 119 | 301
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 3 | 18 | 17 | 1 | 4 | 1 | 6 | 41 | 96
  Male | 4 | 8 | 3 | 7 | 38 | 44 | 4 | 6 | 9 | 4 | 78 | 205
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Bambara | 2 | 5 | 0 | 7 | 14 | 19 | 3 | 5 | 5 | 4 | 27 | 91
  Bozo | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3
  Malinke | 0 | 1 | 2 | 0 | 25 | 24 | 0 | 0 | 2 | 1 | 56 | 111
  Peulh | 0 | 0 | 2 | 1 | 6 | 5 | 1 | 0 | 1 | 1 | 5 | 22
  Sarakole | 0 | 1 | 0 | 1 | 11 | 11 | 0 | 3 | 0 | 3 | 25 | 55
  Sonrhai | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Other | 3 | 3 | 1 | 1 | 0 | 0 | 1 | 2 | 2 | 1 | 3 | 17
Region of Enrollment [Number; unit: participants]
  Mali | 5 | 10 | 5 | 10 | 56 | 61 | 5 | 10 | 10 | 10 | 119 | 301

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Local and Systemic Adverse Events in Year 1
Description: Number of participants with local and systemic adverse events (AEs) graded by severity occurring within 7 days after each vaccine
Time Frame: Within 7 days after each vaccination
Measure: Count of Participants; unit: Participants
Groups:
- Safety/Efficacy Arm 2c: Dosing Interval 0, 28, 168, 476 Days: Participants received 3 doses of 40 μg Pfs230D1M-EPA/AS01 via intramuscular injections into the deltoid muscle (IM) on Days 0, 28, 168, and a 4th dose on Day 476 (Year 2). Participants received antimalarial drug treatment with Coartem® approximately 1 week prior to first vaccination.
  Pfs230D1M-EPA: The Pfs230D1M-EPA was formulated as conjugated Pfs230D1M in 4 mM PBS to a 2X dilution of the high dose (160 (Micro)g/ml in 0.5 ml volume) in cGMP compliance at Walter Reed Bio-production facility in April 2016 and was provided as a single use vial.
  AS01: AS01B adjuvant was provided as a single use vial by GSK, 100 microgram/mL MPL and 100 microgram/mL QS21 in a liposomal formulation in a volume of 0.625 mL. One dose injected of AS01B corresponds to 50 μg QS21 and 50 μg MPL.
  Coartem: Artemether/lumefantrine (Coartem(R)) is a licensed antimalarial in the US and Mali for treatment of uncomplicated malaria. It has an excellent safety profile and is widely used to treat malaria. Subjects who may have had any contraindications to the use of these drugs were excluded at screening. Coartem was dosed with food and administered over 3 days for a total of 6 doses, as per package insert and standard adult dosing
- Pilot/Safety Arm 3a: Dosing Interval 0, 28, 168 Days: Participants received 3 doses of 16 μg Pfs25M-EPA/AS01 and 13 μg Pfs230D1M-EPA/AS01 via intramuscular injections into the deltoid muscle (IM) on Days 0, 28, 168
  Pfs25M-EPA: The PpPfs25M and EcEPA lots, both manufactured at Walter Reed Bioproduction facility (WRB; Silver Spring, Maryland) in cGMP compliance, were used to manufacture the conjugate. PpPfs25M is a Pichia- expressed recombinant Pfs25 with a molecular mass of 18,713 Daltons. The Pfs25M-EPA was formulated as conjugated Pfs25M in 4 mM PBS to a 2X dilution of the high dose (188 μg/ml in 0.5 ml volume) in cGMP compliance at WRB facility in Apr 2016 and provided as a single use vial.
  Pfs230D1M-EPA: The Pfs230D1M-EPA was formulated as conjugated Pfs230D1M in 4 mM PBS to a 2X dilution of the high dose (160 μg/ml in 0.5 ml volume) in cGMP compliance at Walter Reed Bio-production facility in April 2016 and provided as a single use vial.
  AS01: AS01B adjuvant will also be provided as a single use vial by GSK, 100 μg/mL MPL and 100 μg/mL QS21 in a liposomal formulation in a volume of 0.625 mL. One dose injected of AS01B corresponds to 50 μg QS21 and 50 μg MPL.
  Normal Saline: Sterile isotonic (0.9%) normal saline will be commercially procured in the US and shipped to Mali at ambient temperature. Normal saline was administered in a 0.5 mL dose as an intramuscular injection. Normal saline was be used for diluting Pfs25M-EPA and Pfs230D1M-EPA prior to formulation with AS01B for the lower dose groups in Bamako, Mali.
- Pilot/Safety Arm 3b: Dosing Interval 0, 28, 168 Days: Participants received 3 doses of 47 μg Pfs25M-EPA/AS01 and 40 μg Pfs230D1M-EPA/AS01 via intramuscular injections into the deltoid muscle (IM) on Days 0, 28, 168
  Pfs25M-EPA: The PpPfs25M and EcEPA lots, both manufactured at Walter Reed Bioproduction facility (Silver Spring, Maryland) in cGMP compliance, were used to manufacture the conjugate. PpPfs25M is a Pichia-expressed recombinant Pfs25 with a molecular mass of 18,713 Daltons.The Pfs25M-EPA was formulated as conjugated Pfs25M in 4 mM PBS to a 2X dilution of the high dose (188 μg/ml in 0.5 ml volume) in cGMP compliance at Walter Reed Bio-production facility in April 2016 and was provided as a single use vial.
  Pfs230D1M-EPA: The Pfs230D1M-EPA was formulated as conjugated Pfs230D1M in 4 mM PBS to a 2X dilution of the high dose (160 μg/ml in 0.5 ml volume) in cGMP compliance at Walter Reed Bio-production facility in April 2016 and was provided as a single use vial.
  AS01: AS01B adjuvant was provided as a single use vial by GSK, 100 μg/mL MPL and 100 μg/mL QS21 in a liposomal formulation in a volume of 0.625 mL. One dose injected of AS01B corresponds to 50 μg QS21 and 50 μg MPL.
Arm/Group | Pilot/Safety Arm 1a: Dosing Interval 0, 28, 168 Days | Pilot/Safety Arm 1b: Dosing Interval 0, 28, 168 Days | Pilot/Safety Arm 2a: Dosing Interval 0, 28, 168 Days | Pilot/Safety Arm 2b: Dosing Interval 0, 28, 168 Days | Safety/Efficacy Arm 2c: Dosing Interval 0, 28, 168, 476 Days | Safety/Efficacy Arm 2d: Dosing Interval 0, 28, 168, 476 Days | Pilot/Safety Arm 3a: Dosing Interval 0, 28, 168 Days | Pilot/Safety Arm 3b: Dosing Interval 0, 28, 168 Days | Pilot/Safety Comparator Arm 4a: Dosing Interval 0, 28, 168 Days | Pilot/Safety Comparator Arm 4b: Dosing Interval 0, 28, 168 Days | Safety Comparator & Efficacy Comparator Arm 4c: Dosing Interval 0, 28, 168, 476 Days
Number analyzed (Participants) | 5 | 10 | 5 | 10 | 56 | 61 | 5 | 10 | 10 | 10 | 119
Participants | 2 | 6 | 4 | 6 | 31 | 25 | 3 | 8 | 2 | 3 | 52

2. Primary Outcome: Number of Participants With Local and Systemic Adverse Events in Year 2
Description: as for outcome 1
Time Frame: Within 7 days after each vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Safety/Efficacy Arm 2c: Dosing Interval 0, 28, 168, 476 Days | Safety/Efficacy Arm 2d: Dosing Interval 0, 28, 168, 476 Days | Safety Comparator & Efficacy Comparator Arm 4c: Dosing Interval 0, 28, 168, 476 Days
Number analyzed (Participants) | 56 | 61 | 119
Participants | 28 | 27 | 20

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed 7 days from the time of each vaccination in Years 1 and 2
Groups:
- Pilot/Safety Arm 3a: Dosing Interval 0, 28, 168 Days: Participants received 3 doses of 16 μg Pfs25M-EPA/AS01 and 13 μg Pfs230D1M-EPA/AS01 via intramuscular injections into the deltoid muscle (IM) on Days 0, 28, 168
  Pfs25M-EPA: The PpPfs25M and EcEPA lots, both manufactured at Walter Reed Bioproduction facility (WRB; Silver Spring, Maryland) in cGMP compliance, were used to manufacture the conjugate. PpPfs25M is a Pichia- expressed recombinant Pfs25 with a molecular mass of 18,713 Daltons. The Pfs25M-EPA was formulated as conjugated Pfs25M in 4 mM PBS to a 2X dilution of the high dose (188 μg/ml in 0.5 ml volume) in cGMP compliance at WRB facility in April 2016 and was provided as a single use vial.
  Pfs230D1M-EPA: The Pfs230D1M-EPA was formulated as conjugated Pfs230D1M in 4 mM PBS to a 2X dilution of the high dose (160 μg/ml in 0.5 ml volume) in cGMP compliance at WRB facility in April 2016 and was provided as a single use vial.
  AS01: AS01B adjuvant will also be provided as a single use vial by GSK, 100 μg/mL MPL and 100 μg/mL QS21 in a liposomal formulation in a volume of 0.625 mL. One dose injected of AS01B corresponds to 50 μg QS21 and 50 μg MPL.
  Normal Saline: Sterile isotonic (0.9%) normal saline will be commercially procured in the US and shipped to Mali at ambient temperature. Normal saline was administered in a 0.5 mL dose as an intramuscular injection. Normal saline was be used for diluting Pfs25M-EPA and Pfs230D1M-EPA prior to formulation with AS01B for the lower dose groups in Bamako, Mali.
Arm/Group | Pilot/Safety Arm 1a: Dosing Interval 0, 28, 168 Days | Pilot/Safety Arm 1b: Dosing Interval 0, 28, 168 Days | Pilot/Safety Arm 2a: Dosing Interval 0, 28, 168 Days | Pilot/Safety Arm 2b: Dosing Interval 0, 28, 168 Days | Safety/Efficacy Arm 2c: Dosing Interval 0, 28, 168, 476 Days | Safety/Efficacy Arm 2d: Dosing Interval 0, 28, 168, 476 Days | Pilot/Safety Arm 3a: Dosing Interval 0, 28, 168 Days | Pilot/Safety Arm 3b: Dosing Interval 0, 28, 168 Days | Pilot/Safety Comparator Arm 4a: Dosing Interval 0, 28, 168 Days | Pilot/Safety Comparator Arm 4b: Dosing Interval 0, 28, 168 Days | Safety Comparator & Efficacy Comparator Arm 4c: Dosing Interval 0, 28, 168, 476 Days
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/10 | 0/5 | 0/10 | 0/56 | 0/61 | 0/5 | 0/10 | 0/10 | 0/10 | 0/119
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/10 | 0/5 | 0/10 | 0/56 | 0/61 | 0/5 | 0/10 | 0/10 | 1/10 | 1/119
Other Adverse Events (participants affected / at risk) | 2/5 | 7/10 | 5/5 | 8/10 | 53/56 | 58/61 | 4/5 | 9/10 | 4/10 | 4/10 | 79/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot/Safety Arm 1a: Dosing Interval 0, 28, 168 Days (N=5) | Pilot/Safety Arm 1b: Dosing Interval 0, 28, 168 Days (N=10) | Pilot/Safety Arm 2a: Dosing Interval 0, 28, 168 Days (N=5) | Pilot/Safety Arm 2b: Dosing Interval 0, 28, 168 Days (N=10) | Safety/Efficacy Arm 2c: Dosing Interval 0, 28, 168, 476 Days (N=56) | Safety/Efficacy Arm 2d: Dosing Interval 0, 28, 168, 476 Days (N=61) | Pilot/Safety Arm 3a: Dosing Interval 0, 28, 168 Days (N=5) | Pilot/Safety Arm 3b: Dosing Interval 0, 28, 168 Days (N=10) | Pilot/Safety Comparator Arm 4a: Dosing Interval 0, 28, 168 Days (N=10) | Pilot/Safety Comparator Arm 4b: Dosing Interval 0, 28, 168 Days (N=10) | Safety Comparator & Efficacy Comparator Arm 4c: Dosing Interval 0, 28, 168, 476 Days (N=119)
Pulmonary Tuberculosis (Infections and infestations) | NA | NA | NA | NA | NA | NA | NA | NA | NA | 1 (1) | 0
Snake Bite (Injury, poisoning and procedural complications) | NA | NA | NA | NA | NA | NA | NA | NA | NA | 0 | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot/Safety Arm 1a: Dosing Interval 0, 28, 168 Days (N=5) | Pilot/Safety Arm 1b: Dosing Interval 0, 28, 168 Days (N=10) | Pilot/Safety Arm 2a: Dosing Interval 0, 28, 168 Days (N=5) | Pilot/Safety Arm 2b: Dosing Interval 0, 28, 168 Days (N=10) | Safety/Efficacy Arm 2c: Dosing Interval 0, 28, 168, 476 Days (N=56) | Safety/Efficacy Arm 2d: Dosing Interval 0, 28, 168, 476 Days (N=61) | Pilot/Safety Arm 3a: Dosing Interval 0, 28, 168 Days (N=5) | Pilot/Safety Arm 3b: Dosing Interval 0, 28, 168 Days (N=10) | Pilot/Safety Comparator Arm 4a: Dosing Interval 0, 28, 168 Days (N=10) | Pilot/Safety Comparator Arm 4b: Dosing Interval 0, 28, 168 Days (N=10) | Safety Comparator & Efficacy Comparator Arm 4c: Dosing Interval 0, 28, 168, 476 Days (N=119)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 7 (8) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Decreased appetite (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diastolic hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Furuncle (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital infection (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 23 (35) | 25 (29) | 1 (1) | 5 (6) | 1 (1) | 1 (1) | 11 (15)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site movement impairment (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (6) | 2 (2) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 3 (3)
Injection site pain (General disorders) | 2 (3) | 7 (8) | 4 (9) | 7 (13) | 51 (137) | 48 (113) | 4 (12) | 8 (29) | 0 (0) | 3 (3) | 38 (55)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 9 (14)
Malaria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 0 (0) | 3 (5) | 7 (7) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 7 (8)
Oropharyngeal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pharyngitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyoderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (10) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 9 (9)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Systolic hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)

LIMITATIONS AND CAVEATS:
No limitations or caveats to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Before either Party submits a paper or abstract for publication or otherwise intends to publicly disclose information about a CRADA Subject Invention, CRADA Data, or CRADA Materials, the other Party will have thirty (30) days to review proposed manuscripts and fifteen (15) days to review proposed abstracts to assure that Confidential Information is protected.

Dr. Patrick Duffy is employed by the clinical sponsor, NIAID (clinical sponsor). Dr. Sagara is not employed by either sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT02942277/Prot_SAP_000.pdf